CLINICAL TRIAL: NCT02232607
Title: A Randomised, Double-blind, Placebo-controlled, Multi-centre, Parallel Group, Dose Ranging Study to Investigate the Efficacy and Safety of Lacidipine in Chronic Stable Angina.
Brief Title: Efficacy and Safety of Lacidipine in Chronic Stable Angina
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 231.339
Record Dates: First submitted 2014-09-04; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — lacidipine

ARMS (4):
- Lacidipine, low dose (Experimental)
  Interventions: Drug: Lacidipine, low dose; Drug: Placebo
- Lacidipine, medium dose (Experimental)
  Interventions: Drug: Lacidipine, medium dose; Drug: Placebo
- Lacidipine, high dose (Experimental)
  Interventions: Drug: Lacidipine, high dose
- Placebo (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lacidipine, low dose
  Arms: Lacidipine, low dose
Drug: Lacidipine, medium dose
  Arms: Lacidipine, medium dose
Drug: Lacidipine, high dose
  Arms: Lacidipine, high dose
Drug: Placebo
  Arms: Lacidipine, low dose; Lacidipine, medium dose; Placebo

SUMMARY:
The aim of this study was to explore whether lacidipine at doses of 2 mg, 4 mg and 6 mg decreased the symptoms of angina, compared to placebo in patients with chronic stable angina

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* History of stable, exertional angina pectoris (Canadian Cardiovascular Society functional class II to III) for at least 3 months duration prior to enrolment in the study
* Patients not currently receiving treatment with antianginal medication (other than short-acting nitrates)
* Between visits 2 and 3 two treadmill exercise tests, demonstrating ≥ 0.1 mV of horizontal or down sloping ST-segment depression, must be carried out. The difference in symptom-limited exercise duration between these two tests must not exceed 20%
* Total treadmill exercise duration > 3 minutes (i.e. stage 2 or above on a standard Bruce protocol)
* Coronary artery disease, preferably (not mandatory) documented by a history of proven myocardial infarction and/or coronary angiography indicating ≥ 50% reduction in luminal diameter of one or more coronary arteries or their primary branches

Exclusion Criteria:

* Myocardial infarction within 3 months prior to enrolment in the study
* Percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass surgery within 6 months
* Other types of angina (variant, unstable)
* Uncontrolled hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg)
* Resting heart rate < 50 bpm or > 100 bpm
* Significant valvular heart disease
* Heart failure New York Heart Association Class III or IV
* Chronic obstructive pulmonary disease and/or asthma with clinical symptoms requiring regular medication
* Significant arrhythmia (since this may interfere with the interpretation of the electrocardiogram) including Wolff Parkinson-White syndrome, atrial fibrillation, atrial flutter, sick sinus syndrome, significant Atrio-Ventricular heart block, intraventricular conduction defect (QRS > 0.12 seconds) ventricular pre-excitation, bundle branch block, the presence of a pace-maker, the presence of an implanted automatic defibrillator, uncorrected hypokalaemia (potassium < 3.5 mmol/litre)
* Insulin dependent diabetes mellitus
* Significant liver disease (Aspartate Aminotransferase or Alanine Aminotransferase > twice the upper limit of reference range)
* Significant renal disease (creatinine > 1.5 x upper limit of reference range)
* Any clinical condition which in the opinion of the investigator, would preclude the safe fulfilment of the protocol and the safe administration of trial medication
* Inability to perform repeated exercise testing due to extra-cardiac reasons
* Concomitant treatment with any other anti-anginal medication, whether or not prescribed for this indication (e.g. calcium channel blockers, β-blockers or long-acting nitrates)
* Concomitant treatment with anti-arrhythmic medication, digitalis or tricyclic anti-depressants or other agents known to affect ST-segment morphology
* Known hypersensitivity to any of the components of the investigational drug
* Pregnant or nursing women or women of child bearing potential
* Participation in any other clinical trial within 2 months of enrolment
* History of drug or alcohol abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 1998-04; Primary Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
Change in total treadmill exercise duration | Baseline, week 6

SECONDARY OUTCOMES:
Change in time to ST segment depression (≥ 0.1 mV) | up to 6 weeks
Treadmill exercise time to first report of anginal pain | week 6
Reason for termination of treadmill exercise test | up to 6 weeks
Frequency/severity of anginal attacks | up to 6 weeks
Consumption of short-acting nitrates | up to 6 weeks
Number of patients with adverse events | up to 6 weeks